CLINICAL TRIAL: NCT04588532
Title: Characterization of Bovine Adrenal Medulla (BAM8-22) as a New Surrogate Model of Non-histaminergic Itch
Brief Title: Characterization of BAM8-22 as a New Surrogate Model of Non-histaminergic Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Giulia Erica Aliotta, Principal investigator, PhD fellow, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190062 2nd project
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — bovine adrenal medulla 8-22; Histamine; Doxepin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doxepin (Experimental): Drug: Doxepin + BAM8-22 Doxepin will be applied for 1.5 hrs followed by the application of BAM8-22. 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Doxepin + Histamine Doxepin will be applied for 1.5 hrs followed by the application of Histamine. 20 µl of histamine will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Doxepin + Cowhage Doxepin will be applied for 1.5 hrs followed by the application of cowhage. 25/35 spicules of cowhage will be inserted in the skin through a gentle rubbing on a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Doxepin + Placebo Doxepin will be applied for 1.5 hrs followed by the application of placebo. 20 µl of placebo will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Interventions: Drug: BAM8-22; Drug: Histamine; Drug: Cowhage (Mucuna Pruriens); Drug: Doxepin
- itch (Experimental): Drug: BAM8-22 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Histamine 20 µl of histamine will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Cowhage 25/35 spicules of cowhage will be inserted in the skin through a gentle rubbing on a previously determined area on the volar forearm followed by a prick through the drop
  Drug: Placebo 20 µl of placebo will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Interventions: Drug: BAM8-22; Drug: Histamine; Drug: Cowhage (Mucuna Pruriens)

INTERVENTIONS:
Drug: BAM8-22 — Bovine Adrenal Medulla will be applied to 2 previously determined area on the volar forearm (one alone and one in combination with doxepin)
Drug: Histamine — histamine will be applied to 2 previously determined area on the volar forearm (one alone and one in combination with doxepin)
Drug: Cowhage (Mucuna Pruriens) — cowhage spicules will be applied to 2 previously determined area on the volar forearm (one alone and one in combination with doxepin)
Drug: Doxepin — Doxepin cream (antihistamine) will be applied in 4 areas on the volar forearm
  Arms: doxepin

SUMMARY:
With this experiment, the experimenter wish to asses if substance BAM8-22 (Bovine Adrenal Medulla) induce non-histaminergic itch.

DETAILED DESCRIPTION:
With this experiment, the experimenter wish to establish if the substance BAM8-22 (Bovine Adrenal Medulla) induce a non-histaminergic itch by using the antihistamine Doxepin.

The experimenter will also compare itch and the response to antihistamine of BAM8-22, histamine and cowhage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.)
* Moles, wounds, scars or tattoos in the area to be treated or tested
* Lack of ability to cooperate •
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these - Acute or chronic pain •
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
superficial blood perfusion | change from baseline, up to 10 minutes after the first session
  is measured by a speckle contrast imager (FLPI, Moor Instruments, England)
Warm Detection Threshold, and Heat Pain threshold | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Threshold and Cold Pain threshold | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain supra-threshold heat Stimuli | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
hyperknesis (abnormal pruriceptive state) | change from baseline, up to 10 minutes after the first session
  is measured by using a mildly pruritic, non-painful von Frey filaments of a predetermined intensity (generally 5-30 milliNewton of force)
mechanical pain threshold and sensitivity | change from baseline, up to 10 minutes after the first session
  is performed using a pin-prick set (Aalborg University). The set consists of 8 needles each having a diameter of 0,6 mm and different force applications
itch rating | change from baseline, up to 10 minutes after the first session
  the subject will rate the itch for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no itch" and 100 indicates "worst imaginable itch"

SECONDARY OUTCOMES:
pain rating | change from baseline, up to 10 minutes after the first session
  the subject will rate the pain for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no pain" and 100 indicates "worst imaginable pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark